CLINICAL TRIAL: NCT01739829
Title: A Phase I/IIa Open-label Investigation of the Safety and Effectiveness of DIABECELL® [Immunoprotected (Alginate-Encapsulated) Porcine Islets for Xenotransplantation] in Patients With Type 1 Diabetes Mellitus
Brief Title: Open-label Investigation of the Safety and Effectiveness of DIABECELL® in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diatranz Otsuka Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCT/DIA-09
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes
Keywords: xenotransplantation; type 1 diabetes; porcine islets
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DIABECELL group 1 (Experimental): 10,000 IEQ per kg body weight (Total Dose) Administered in two doses: 5,000 IEQ/kg three months apart.
  Interventions: Device: DIABECELL (R)
- DIABECELL group 2 (Experimental): 20,000 IEQ per kg body weight (Total Dose) Administered in two doses: 10,000 IEQ/kg three months apart
  Interventions: Device: DIABECELL (R)

INTERVENTIONS:
Device: DIABECELL (R) — 10,000 IEQ per kg body weight (Total Dose) Administered in two doses: 5,000 IEQ/kg three months apart.
  Arms: DIABECELL group 1
Device: DIABECELL (R) — 20,000 IEQ per kg body weight (Total Dose) Administered in two doses: 10,000 IEQ/kg three months apart
  Arms: DIABECELL group 2

SUMMARY:
The purpose of this study is to establish the safety and efficacy of xenotransplantation of DIABECELL® in patients with established type 1 diabetes mellitus

DETAILED DESCRIPTION:
Intraperitoneal islet transplantation has the potential to ameliorate type 1 diabetes mellitus and avert the long-term consequences of chronic diabetes which cannot be achieved by conventional insulin treatment.

As donor human islets are not available in sufficient numbers, porcine islets are the best alternative source as they are recognised as the most physiologically compatible xenogeneic insulin-producing cells. Although the use of pig-derived cells raises the risk of xenotic infections, this can be minimised by obtaining cells from designated pathogen-free (DPF) animals bred in isolation and monitored to be free of specified pathogens. The worldwide experience to date in more than 200 patients who have received transplants of pig tissue has not demonstrated evidence of transmitted xenotic infections.

As animal-derived tissues have to be protected from immune rejection when transplanted into humans, transplants are usually accompanied by immunosuppressive therapy. However, porcine islets are preferably transplanted without the use of immunosuppressive drugs which cause significant morbidity. To protect them from immune rejection, the islets can be encapsulated in alginate microcapsules which permit the inward passage of nutrients and glucose and the outward passage of insulin. Alginate-encapsulated porcine islets transplanted without immunosuppressive drugs have survived rejection for many months in animal studies, and have been retrieved from a diabetic patient over 9.5 years after intraperitoneal transplantation and shown to contain viable islets that stain positive for insulin.

DIABECELL® comprises neonatal porcine islets encapsulated in alginate microcapsules. DIABECELL® has been safely transplanted in healthy and diabetic mice, rats, rabbits, dogs and non-human primates. Following DIABECELL® transplants, the requirement for daily insulin was significantly reduced in diabetic rats and non-human primates.

The optimal dose and frequency of transplantation of the current DIABECELL® preparation for the treatment of type 1 diabetes in humans can only be determined in clinical trials. The intention of this phase I/IIa clinical trial is to obtain at least 52 weeks safety and preliminary efficacy data in type 1 diabetic patients following transplantation of two low effective doses of DIABECELL® into the peritoneal cavity.

ELIGIBILITY:
Inclusion Criteria:

Adults (males or females) in the age range 18 to 65 years

* Diagnosis of type 1 diabetes mellitus (minimum duration of 5 years) in accordance with the American Diabetes Association's criteria. Patients should have been treated continuously with insulin since diagnosis (Expert Committee on the Diagnosis and Classification of Diabetes Mellitus 2002)
* Patients with established brittle type I diabetes mellitus with a well-documented chronic history of metabolic instability who cannot achieve acceptable metabolic control (which may include treatment with the use of a continuous insulin infusion pump) without experiencing multiple episodes of hypoglycaemia, often with unawareness
* Patients should have an HbA1C ≥7% and ≤15% calculated as the average of the last four consecutive HbA1C readings during the 8-week baseline run-in period. The difference between the highest and lowest of the four HbA1C reading should be no more than 1.0%.
* Plasma C-peptide <0.3 ng/ml following a glucagon stimulation test (Scheen et al. 1996)
* If female, no childbearing capability (those who are more than two years post menopausal or have undergone voluntary sterilisation can be considered for enrolment)
* Provision of written informed consent. Patients will be required to agree to comply with all tests and visits specified in the protocol, and they (and their partners/close contacts) will also be required to consent to long-term microbiological monitoring, which is an integral part of the study

Exclusion Criteria:

* Type 2 diabetes, defined as age of onset >30 years and/or a history of treatment with oral hypoglycaemic medications and/or insulin resistance (defined as an insulin dose requirement ≥1.2 U/kg/day)
* An average HbA1C < 7% and >15% during the 8-week baseline run-in period
* Body mass index (BMI) ≥30 kg/m2 or ≤9 kg/m2
* Active infection, with plasma C-reactive protein ≥10 mg/L at baseline
* Previous receipt of an organ, skin graft, or other tissue transplant from a human or animal donor
* Treatment with immunosuppressive medications for another medical condition
* Previous history of peritoneal disease or abnormal findings at baseline laparoscopy
* Previous abdominal surgery, excluding uncomplicated appendectomy, cholecystectomy or caesarean section
* History of pelvic inflammatory disease or endometriosis
* Inability to tolerate oral medications or a history of significant malabsorption
* HIV antibody and/or risk factors for HIV infection
* Positive hepatitis C antibody, positive hepatitis B surface antigen and hepatitis B core antibody
* Kidney disease, defined as serum creatinine >130 μmol/L in men and >110 μmol/L in women and/or urinary albumin >500 mg/L and/or haematuria and/or active urinary sediment or casts
* Diabetes microvascular complications defined as untreated, potentially vision-threatening proliferative or pre-proliferative retinopathy or maculopathy; painful peripheral neuropathy; autonomic neuropathy manifesting as postural hypotension; gastroparesis or diabetic enteropathy
* Diagnosis of coeliac disease and history of gastrointestinal symptoms including chronic or recurrent diarrhoea, malabsorption, weight loss and abdominal distension or bloating on exposure to gluten products in the diet
* Serious comorbid conditions that are likely to affect participation in the study, including:

  1. Previous coronary heart disease manifesting as non-ST elevation myocardial infarction (NSTEMI), Q-wave infarction or unstable angina; coronary artery bypass graft (CABG); or percutaneous angioplasty
  2. Previous cerebrovascular disease manifesting as transient ischaemic attacks (TIAs) or stroke
  3. Peripheral vascular disease with previous amputation
  4. History of New York Heart Association (NYHA) class II, III or IV congestive heart failure (CHF) and/or chronic atrial fibrillation
  5. Chronic obstructive pulmonary disease (COPD) or asthma with previous hospitalisation for decompensation; a requirement for mechanical ventilation at any stage; or long-term treatment with oral corticosteroids
  6. Liver disease with abnormal liver function tests defined as serum bilirubin ≥20 µmol/L, and/or ALT ≥100 U/L, and/or GGT ≥100 U/L, and/or albumin <35 g/L
  7. Haematological disorders, including haemoglobin ≤110 g/L or platelet count <80 x 109/L
  8. Peptic ulcer disease and/or history of previous gastrointestinal bleeding
  9. Malignancy other than basal cell carcinoma
  10. History of epilepsy
  11. Untreated hypothyroidism
  12. Known adrenal insufficiency
* History of drug, substance or alcohol addiction
* Any factor detected from psychometric evaluation at Visit 2 Pre-Tx during the screening period which may in the opinion of the Clinical Psychologist affect an individual's ability to fully participate in the study
* Any other condition that, in the opinion of the Investigator, may interfere with adherence to the study protocol, including dementia, mental illness, or a history of non-adherence to appointments or treatments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To establish the safety and efficacy of xenotransplantation of DIABECELL | 2 years
  * safety determined by occurence of hypoglycaemic events, occurence of perioperative reactions, occurence of adverse/serious adverse events, monitoring laboratory test results (including xenogeneic infection status), conducting physical examination, ECG
  * efficacy determined by change in HbA1c,daily insulin dose, transplant estimate function score, time spent in euglycaemia, occurence of hypoglycaemic events, quality of life assessment
  * the primary endpoint will be a reduction in the unaware hypoglycaemic event rate combined with no increase in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Abalovich, Principal Investigator — Eva Perón Hospital, San Martín
Locations (1):
- Hospital Interzonal General de Agudos Eva Perón, Buenos Aires, Argentina

REFERENCES:
- See also: Diatranz Otsuka Limited — http://www.dolglobal.com/